CLINICAL TRIAL: NCT00710970
Title: H-16848 - Phase II Pilot Study With Correlative Markers of Tamoxifen for Progressive Transitional Cell Carcinoma Following Previous Chemotherapy
Brief Title: Tamoxifen for Progressive Transitional Cell Carcinoma Following Previous Chemotherapy Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seth Lerner (Other)
Collaborators: AstraZeneca (Industry); Cytogen Corporation (Industry)
Responsible Party: Sponsor-Investigator, Seth Lerner, Professor, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-16848; NCT00589017 (obsolete NCT alias)
Record Dates: First submitted 2008-07-07; First posted 2008-07-08 (Estimated); Results first posted 2013-08-22 (Estimated); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: Urinary Bladder Neoplasms
Keywords: Urinary Bladder Neoplasms; Previous Chemotherapy; Tamoxifen; Anti-tumor activity
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Tamoxifen; Raloxifene Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm Receiving 25mg Tamoxifen (Experimental)
  Interventions: Drug: Tamoxifen

INTERVENTIONS:
Drug: Tamoxifen — Tamoxifen is administered at 20 mg/day as a single daily oral dose. Tamoxifen is continued until progressive disease or intolerable grade 3 or 4 side effects occur due to tamoxifen.
  Other Names: raloxifene

SUMMARY:
The major objective of this two-stage phase II study is to determine whether tamoxifen is deserving of further study in metastatic bladder cancer. Tamoxifen is expected to function as a cytostatic (and not cytotoxic) agent, and may produce more disease stability than regression. Sustained stable disease is considered to be clinically important and the more likely event. Hence, 4-month freedom from progression is chosen as the primary end-point instead of response rate. Freedom from progression is defined as the period from start of therapy to the time of objective radiologic progression. A total of 25 subjects will be enrolled, 15 during stage 1 and 10 during stage 2 of a two-stage minimax design phase II study.

Pre-therapy evaluation (within 3 weeks of initiation of therapy):

* History and physical examination (H and P)
* Performance status (PS) assessment
* CBC (complete blood counts)
* CMP (complete metabolic profile)
* Pregnancy test (in women younger than 50)
* Computed tomography (CT) scan of the chest, abdomen and pelvis
* Bone scan if bone pain or raised alkaline phosphatase
* Biopsy (may use previous biopsy specimen)
* Samples of plasma from the routine CBC and CMP will be banked indefinitely for future biomarker studies at the Scott Department of Urology.

Treatment plan: Therapy will be administered as an outpatient. Tamoxifen is administered at 20 mg/day as a single daily oral dose. Clinical assessment of patients by a history and physical examination will be performed every 4 weeks (one cycle). Objective radiological assessment of response will be made every 8 weeks or earlier if clinically indicated. A CT (computerized tomography) scan of the abdomen, pelvis and chest will be performed at baseline and every 2 cycles. A response is confirmed by repeating the scans in 4 weeks. Bone scan is performed if the patient complains of new bone pain or has raised alkaline phosphatase. A radiologist who is blinded to the treatment regimen reads the scans. The RECIST criteria are used to define response. Tamoxifen is continued until progressive disease or intolerable side effects occur.

ELIGIBILITY:
Inclusion Criteria:

* Patients previously diagnosed with bladder cancer who have already received 1-2 systemic therapy regimens (chemotherapy or biological therapy or both) but including at least one chemotherapy regimen.
* Patients who have had the cancer spread to other parts of the body.
* Patients must have adequate liver function.

Exclusion Criteria:

* Patients who have uncontrolled nervous system metastasis
* Patients who are pregnant
* Patients who have had systemic therapies within the past 4 weeks
* Patients who plan to have major surgery within 2 weeks
* Patients who have Grade III/IV heart problems
* Patients who have severe and/or uncontrolled medical disease.
* Patients who might be at high risk for deep vein thrombosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2007-01; Primary Completion 2011-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seth P. Lerner, M.D., Principal Investigator — Baylor College of Medicine
Locations (2):
- Baylor College Of Medicine, Houston, Texas, United States
- San Camillo and Forlanini Hospitals, Rome, Italy

REFERENCES:
- [Background] Kim HT, Kim BC, Kim IY, Mamura M, Seong DH, Jang JJ, Kim SJ. Raloxifene, a mixed estrogen agonist/antagonist, induces apoptosis through cleavage of BAD in TSU-PR1 human cancer cells. J Biol Chem. 2002 Sep 6;277(36):32510-5. doi: 10.1074/jbc.M202852200. Epub 2002 Jun 25. PMID 12084714
- [Background] Shen SS, Smith CL, Hsieh JT, Yu J, Kim IY, Jian W, Sonpavde G, Ayala GE, Younes M, Lerner SP. Expression of estrogen receptors-alpha and -beta in bladder cancer cell lines and human bladder tumor tissue. Cancer. 2006 Jun 15;106(12):2610-6. doi: 10.1002/cncr.21945. PMID 16700038
- See also: Baylor College of Medicine's Clinical Trials — http://www.bcm.edu/clinicalstudies
- See also: Scott Department of Urology, Baylor College of Medicine — http://www.baylorurology.org
- See also: Bladder Cancer Advocacy Network — http://bcan.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients presenting to the Scott Department of Urology for management of recurrent bladder cancer and fulfill the following criteria will be recruited.
Groups:
- Single Arm Receiving 20mg Tamoxifen: Tamoxifen : Tamoxifen is administered at 20 mg/day as a single daily oral dose. Tamoxifen is continued until progressive disease or intolerable grade 3 or 4 side effects occur due to tamoxifen.
Period: Overall Study
Arm/Group | Single Arm Receiving 20mg Tamoxifen
Started | 28
Completed | 25
Not Completed | 3
Not completed — Never took drug | 3

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm Receiving 20mg Tamoxifen
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (10.844)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 26
Region of Enrollment [Number; unit: participants]
  United States | 21
  Italy | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Freedom From Progression of Cancer at 4 Months
Description: Clinical Assessments were performed every 4 weeks and imaging every 8 weeks or earlier if indicated.
  Patients were followed every month for clinical symptoms and signs of progression.
  Patients underwent Radiographic CT scans every 8 weeks to look for progression.
Time Frame: Estimated from date of starting therapy until 4 months but up to progression or death which ever comes first.
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm Receiving 25mg Tamoxifen
Number analyzed (Participants) | 20
Participants | 20

ADVERSE EVENTS:
Arm/Group | Single Arm Receiving 20mg Tamoxifen
Serious Adverse Events (participants affected / at risk) | 2/19
Other Adverse Events (participants affected / at risk) | 18/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm Receiving 20mg Tamoxifen (N=19)
Acute Renal Failure (Renal and urinary disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 2.8% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm Receiving 20mg Tamoxifen (N=19)
Allergic Rhinitis (Immune system disorders) | 1
anemia (Blood and lymphatic system disorders) | 6
Decreased hematocrit (Blood and lymphatic system disorders) | 5
Decreased hemoglobin (Blood and lymphatic system disorders) | 4
Decreased lymphocytes (Blood and lymphatic system disorders) | 4
Decreased Red Blood Cells (Blood and lymphatic system disorders) | 1
Decreased White Blood Cells (Blood and lymphatic system disorders) | 1
Increased Granulocytes (Blood and lymphatic system disorders) | 1
Increased Monocytes (Blood and lymphatic system disorders) | 1
Increased neutrophil (Blood and lymphatic system disorders) | 1
Increased White Blood Cell (Blood and lymphatic system disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Chest Pain (Blood and lymphatic system disorders) | 1
Hypertension (Cardiac disorders) | 1
Hypotension (Cardiac disorders) | 1
Fatigue (Investigations) | 4
Hot Flashes (Endocrine disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Flatuence (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Vomitting (Gastrointestinal disorders) | 1
Anorexia (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Sepsis (Infections and infestations) | 1
Sinus Infection (Infections and infestations) | 1
Decreased Alk Phos (Metabolism and nutrition disorders) | 1
Decreased ALT (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 3
Increased Albumin (Metabolism and nutrition disorders) | 1
Increased Alk Phos (Metabolism and nutrition disorders) | 5
Increased Bilirubin (Metabolism and nutrition disorders) | 1
Increased BUN (Investigations) | 3
Increased Creatinine (Investigations) | 6
Increased ferritin (Investigations) | 1
Increased SGOT (Investigations) | 3
Dizziness (Nervous system disorders) | 4
Neuropathy (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Pain in Anus (General disorders) | 1
Pain in upper thigh (General disorders) | 1
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Hematuria (Renal and urinary disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Pyleonephritis (Renal and urinary disorders) | 1
Cellulitis (Infections and infestations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No